CLINICAL TRIAL: NCT00511875
Title: Evaluation of Effect of Doxycycline Verses Placebo on Diabetic Retinopathy Progression and Retinal Function in Patients With Severe Non-proliferative or Mild or Moderate (Non-high-risk) Proliferative Diabetic Retinopathy
Brief Title: Evaluation of Doxycycline Verses Placebo for the Treatment of Severe Nonproliferative or Mild or Moderate Proliferative Diabetic Retinopathy
Acronym: POC1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Thomas Gardner (Other)
Collaborators: Juvenile Diabetes Research Foundation (Other)
Responsible Party: Sponsor-Investigator, Thomas Gardner, Thomas W. Gardner, MD, Milton S. Hershey Medical Center
Organization: Milton S. Hershey Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 25234; EudraCT number: 2007-005601-22
Record Dates: First submitted 2007-08-03; First posted 2007-08-06 (Estimated); Results first posted 2018-11-02 (Actual); Last update posted 2018-11-02 (Actual); Status verified 2018-10

CONDITIONS: Diabetic Retinopathy
Keywords: diabetic retinopathy; diabetes; diabetic eye studies; neovascularization
MeSH Terms: conditions — Diabetic Retinopathy; Diabetes Mellitus; Neovascularization, Pathologic | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Doxycycline Monohydrate (Experimental): stratified equally to doxycycline monohydrate 50mg taken once daily for 24 months
  Interventions: Drug: doxycycline monohydrate
- Placebo (Placebo Comparator): stratified equally to placebo taken once daily for 24 months
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: doxycycline monohydrate — 50mg once daily for 24 months
  Other Names: doxycycline
  Arms: Doxycycline Monohydrate
Drug: placebo — placebo taken once daily for 24 months
  Arms: Placebo

SUMMARY:
This 24 month randomized research study will evaluate whether doxycycline can 1) slow the deterioration or improve retinal function and/or 2) induce regression, or slow progression, of diabetic retinopathy in participants over 18 years of age with type 1 or type 2 diabetes with severe non-proliferative or early proliferative diabetic retinopathy.

DETAILED DESCRIPTION:
The objectives of this proof-of-concept study are to investigate whether doxycycline can 1) slow the deterioration or improve retinal function and/or 2) induce regression, or slow progression, of diabetic retinopathy. The tests will be performed in the Ophthalmology Departments of the Penn State College of Medicine and Glostrup Hospital, Copenhagen, Denmark. The 24 month proof-of-concept clinical study will involve a prospective, randomized, double-masked clinical trial including 60 adult patients with type 1 or type 2 diabetes who have severe non-proliferative diabetic retinopathy (ETDRS level 53E) or mild or moderate proliferative diabetic retinopathy (retinal and /or optic disk neovascularization less than the "high-risk" ETDRS level 61 or 65), neovascularization of the disc or neovascularization elsewhere >1/2 disc area and in whom panretinal photocoagulation is not imminently required in the ophthalmologist's judgment.

Systemic Exclusion Criteria:

* unstable medical status (e.g. glycemic control, blood pressure, cardiovascular disease) in the opinion of investigator
* significant renal disease (defined as a serum creatinine > 2.5 mg/dL),
* systolic blood pressure > 180 mm Hg or diastolic blood pressure > 110 mm Hg
* history of headaches associated with tetracycline therapy
* history of pseudotumor cerebri
* pregnancy; for women of child-bearing potential, a serum pregnancy test will be performed.
* lactating or intending to become pregnant during the study period (at least 24 months)
* sexually active women of child-bearing potential not actively practicing birth control by using a medically accepted device or therapy (that is, intrauterine device, hormonal contraceptive, or barrier devices) during the study period (at least 24 months); since doxycycline may interfere with the effectiveness of hormonal contraceptives, sexually active women of child-bearing potential who use a hormonal contraceptive will be required to use a second form of contraception to safeguard against contraceptive failure while participating in the study
* known allergy/intolerance to doxycycline or any ingredient in the study drug or placebo (e.g. cellulose, hypromellose, iron oxide, methacrylic acid copolymer, polyethylene glycol, polysorbate 80, sugar spheres, talc, titanium dioxide, and triethyl citrate)
* patients taking phenytoin, barbiturates or carbamazepine, with gastroparesis, with a history of gastrectomy, gastric bypass surgery or otherwise deemed achlorhydric or with a BMI > 30 kg/m2 will also be excluded because of altered doxycycline pharmacokinetics and/or bioavailability
* patients taking strontium, acitretin or tretinoin will be excluded due to the potential for serious drug interactions with doxycycline
* patients with abnormal ALT or AST at baseline will be referred to their primary care physician for medical clearance for participation in this study

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old
* diagnosis of type 1 or type 2 diabetes mellitus
* have a hemoglobin A1c less than 11% at pre-qualification visit
* able and willing to give informed consent
* best-corrected ETDRS visual acuity in study eye ≥ 49 letters (20/100)
* severe non-proliferative diabetic retinopathy (ETDRS level 53E) or retinal and/or optic disk neovascularization less than the "high-risk" characteristics defined by the Diabetic Retinopathy Study (ETDRS level61- 65), and in whom panretinal photocoagulation is not imminently required in the ophthalmologist's judgment
* able to perform reliable visual field and dark adaptation testing
* central subfield thickness on OCT of ≤ 275microns
* foveal fixation present in each eye (assessed by fundus photography using an internal fixation pointer or assessed by the investigator)
* media clarity and pupil dilation sufficient for high-quality fundus photographs and fluorescein angiograms

Exclusion Criteria:

* high-risk neovascularization in study eye
* prior panretinal photocoagulation in the study eye
* focal/grid laser photocoagulation in the macula within the past 15 weeks in the study eye
* intraocular pressure > 22mmHg by Goldmann Tonometry in the study eye
* history of pars plana vitrectomy in the study eye
* vitreous or pre-retinal hemorrhage in the study eye
* systemic or intravitreal anti-VEGF agent to the study eye or the fellow eye within the past 3 months
* peribulbar steroid injection to the study eye or the fellow eye within the past 6 months
* intravitreal triamcinolone acetonide to the study eye within the past 4 months
* expectation by the investigator that retinal photocoagulation or other treatment for diabetic retinopathy (e.g. focal/grid laser to study eye, intravitreal triamcinolone acetonide to study eye, intravitreal anti-VEGF agent to study or fellow eye, ruboxistaurin or systemic anti-VEGF agent for diabetic macular edema) will be administered in the subsequent 24 months
* an ocular condition (other than diabetes) is present in the study eye that, in the opinion of the investigator, might alter visual acuity during the course of the study (e.g. retinal vein occlusion, uveitis or other ocular inflammatory disease, neovascular glaucoma, Irvine-Gass Syndrome, etc)
* anticipated need for cataract surgery in the study eye in the subsequent 24 months in the opinion of the investigator
* history of major ocular surgery (including cataract surgery, scleral buckle, any intraocular surgery, etc) in the study eye within prior 6 months or anticipated within the subsequent 24 months following randomization
* aphakia in the study eye
* history of YAG capsulotomy performed in the study eye within 2 months prior to randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2008-07; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thomas W Gardner, MD MS, Study Director — University of Michigan, Kellogg Eye Center
Locations (1):
- Penn State College of Medicine, Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania, United States

REFERENCES:
- [Derived] Scott IU, Jackson GR, Quillen DA, Larsen M, Klein R, Liao J, Holfort S, Munch IC, Gardner TW. Effect of doxycycline vs placebo on retinal function and diabetic retinopathy progression in patients with severe nonproliferative or non-high-risk proliferative diabetic retinopathy: a randomized clinical trial. JAMA Ophthalmol. 2014 May;132(5):535-43. doi: 10.1001/jamaophthalmol.2014.93. PMID 24604308
- See also: Penn State University, Milton S. Hershey Medical Center — http://www.hmc.psu.edu
- See also: Juvenile Diabetes Research Foundation — http://jdrf.org
- See also: Penn State Hershey Eye Center, Department of Ophthalmology — http://www.pennstatehershey.org/web/eyecenter/home

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Doxycycline Monohydrate | Placebo
Started | 15 | 15
Completed | 10 | 15
Not Completed | 5 | 0
Not completed — Lost to Follow-up | 4 | 0
Not completed — Missing variables | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Doxycycline Monohydrate | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 9 | 12 | 21
  >=65 years | 6 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 9 | 9 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 15 | 12 | 27
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 6 | 8 | 14
  Denmark | 9 | 7 | 16

OUTCOME MEASURES:

1. Primary Outcome: Change in Dark Adaptation, Rod Intercept
Description: Change in dark adaptation is measured as dark adaptation time at baseline measured in minutes minus dark adaptation time measured at 24 months
Time Frame: Baseline and 24 months
Population: Of 10 participants who completed doxycycline treatment, usable endpoint data is only available for 8.
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 8
minutes | 0.3 (3.3) | -0.3 (3.2)
Statistical Analysis 1: Comparison: Placebo vs Doxycycline Monohydrate; Test type: Superiority; p = .70, t-test, 2 sided

2. Primary Outcome: Change in Photopic Visual Field
Description: Change in photopic visual fields between baseline and 24 months
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 10
dB
  Foveal Sensitivity | -0.8 (12.2) | -0.8 (1.3)
  Mean Sensitivity | -0.74 (1.90) | -1.0 (2.4)
Statistical Analysis 1: Comparison: Placebo vs Doxycycline Monohydrate; Foveal Sensitivity; Test type: Superiority; p = .33, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Doxycycline Monohydrate; Mean field sensitivity; Test type: Superiority; p = .16, t-test, 2 sided

3. Primary Outcome: Change in Frequency Doubling Perimetry (FDP)
Description: Change in Frequency Doubling Perimetry (FDP) from baseline, shown as mean and foveal (center of retina) scores
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 10
dB
  Foveal Sensitivity | -1.9 (3.8) | 1.8 (3.6)
  Mean FDP sensitivity | -0.7 (3.9) | 0.7 (2.7)
Statistical Analysis 1: Comparison: Placebo vs Doxycycline Monohydrate; Foveal Sensitivity; Test type: Superiority; p = .02, t-test, 2 sided
Statistical Analysis 2: Comparison: Placebo vs Doxycycline Monohydrate; mean FDP sensitivity; Test type: Superiority; p = .3, t-test, 2 sided

4. Primary Outcome: Change in Early Treatment Diabetic Retinopathy Study (ETDRS)
Description: Change in ETDRS visual acuity letter score from baseline. ETDRS is measured on a scale of 0 to 70 where 0 means inability to see anything on the chart and 70 is normal (20/20) acuity.
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 11
score on a scale | 0.3 (8.8) | 0.2 (4.9)
Statistical Analysis 1: Comparison: Placebo vs Doxycycline Monohydrate; Test type: Superiority; p = .98, t-test, 2 sided

5. Secondary Outcome: Change in Central Subfield Thickness
Description: Change in central subfield thickness from baseline
Time Frame: Baseline and 24 months
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 11
μm | -1.5 (14.9) | 4.8 (26.3)
Statistical Analysis 1: Comparison: Placebo vs Doxycycline Monohydrate; Test type: Superiority; p = .46, t-test, 2 sided

6. Secondary Outcome: Change in Macular Volume
Description: Change in macular volume from baseline
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: mm^3
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 11
mm^3 | -0.2 (0.3) | -0.1 (0.7)
Statistical Analysis 1: Comparison: Placebo vs Doxycycline Monohydrate; Test type: Superiority; p = .81, t-test, 2 sided

7. Secondary Outcome: Change in Central Retinal Artery Equivalent (CRAE) Diameter
Description: Change in Central Retinal Artery Equivalent (CRAE) diameter from baseline
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 11
μm | -0.49 (12) | 0.17 (14)
Statistical Analysis 1: Comparison: Placebo vs Doxycycline Monohydrate; Test type: Superiority; p = .88, t-test, 2 sided

8. Secondary Outcome: Change in Central Retinal Vein Equivalent (CRVE) Diameter
Description: Change in Central Retinal Vein Equivalent (CRVE) diameter from baseline
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: μm
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 11
μm | -6.3 (19) | -6.6 (18)
Statistical Analysis 1: Comparison: Placebo vs Doxycycline Monohydrate; Test type: Superiority; p = .75, t-test, 2 sided

9. Secondary Outcome: Change in Arteriovenous Ratio Diameter
Description: Change in arteriovenous ratio diameter from baseline
Time Frame: 24 months
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Placebo | Doxycycline Monohydrate
Number analyzed (Participants) | 15 | 11
ratio | 0.013 (0.057) | 0.013 (0.056)
Statistical Analysis 1: Comparison: Placebo vs Doxycycline Monohydrate; Test type: Superiority; p = .62, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | Placebo | Doxycycline Monohydrate
Serious Adverse Events (participants affected / at risk) | 3/15 | 3/15
Other Adverse Events (participants affected / at risk) | 14/15 | 15/15
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Doxycycline Monohydrate (N=15)
motor vehicle accident (Injury, poisoning and procedural complications) | 1 | 0
elevated serum creatinine level (Blood and lymphatic system disorders) | 1 | 0
persistent vitreous hemorrhage (Eye disorders) | 0 | 1
pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
concussion of brain (Nervous system disorders) | 1 | 0
umbilical hernia (Gastrointestinal disorders) | 0 | 1
vomiting (Gastrointestinal disorders) | 0 | 1
skull fracture (Injury, poisoning and procedural complications) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=15) | Doxycycline Monohydrate (N=15)
abscess molar tooth (root canal) (Musculoskeletal and connective tissue disorders) | 1 | 0
allergic reaction - reason unknown (Immune system disorders) | 1 | 0
allergies (seasonal) (Immune system disorders) | 1 | 0
ankle sprain (right) (Musculoskeletal and connective tissue disorders) | 1 | 0
anxiety (mild) (Psychiatric disorders) | 1 | 1
back pain (possibly with neck pain) (Musculoskeletal and connective tissue disorders) | 2 | 2
benign prostatic hyperplasia (Renal and urinary disorders) | 1 | 0
bilateral blepharitis (Skin and subcutaneous tissue disorders) | 3 | 0
broken right foot (Injury, poisoning and procedural complications) | 1 | 0
bronchitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
burning sensation in fingers (Nervous system disorders) | 1 | 0
carpal tunnel surgery (left) (Surgical and medical procedures) | 0 | 1
cataract (Eye disorders) | 1 | 0
cataract extraction (Surgical and medical procedures) | 1 | 0
chalazion left eye (Eye disorders) | 0 | 1
chest cold (Respiratory, thoracic and mediastinal disorders) | 0 | 2
congestive heart failure (Cardiac disorders) | 1 | 0
constipation (Gastrointestinal disorders) | 0 | 1
cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1
decreased smell (Nervous system disorders) | 1 | 0
decreased taste (Nervous system disorders) | 1 | 0
depression (Psychiatric disorders) | 1 | 0
diarrhea (Gastrointestinal disorders) | 1 | 0
diplopia (Eye disorders) | 1 | 0
dry rash (Skin and subcutaneous tissue disorders) | 0 | 1
epidermoid cyst (Skin and subcutaneous tissue disorders) | 0 | 1
epiretinal fibrosis (Eye disorders) | 1 | 1
epiretinal membrane, (slight) right eye (Eye disorders) | 0 | 1
fall (cause of injuries unknown) (Injury, poisoning and procedural complications) | 0 | 2
fatigue (General disorders) | 0 | 1
flashes right eye (Eye disorders) | 1 | 0
floaters left eye (Eye disorders) | 1 | 0
flu (Infections and infestations) | 4 | 1
fluid on left knee (Musculoskeletal and connective tissue disorders) | 0 | 1
gastric ulcer (Gastrointestinal disorders) | 1 | 0
gout (Metabolism and nutrition disorders) | 0 | 1
head cold (Respiratory, thoracic and mediastinal disorders) | 0 | 1
headaches (Nervous system disorders) | 1 | 2
high creatinine (Renal and urinary disorders) | 2 | 2
high intraocular pressure (Eye disorders) | 1 | 0
high urine albumin (Renal and urinary disorders) | 1 | 0
hyperlipidemia (Metabolism and nutrition disorders) | 1 | 0
hypertension (Cardiac disorders) | 4 | 1
hypoglycemic episode (Metabolism and nutrition disorders) | 3 | 0
impacted wisdom tooth (Musculoskeletal and connective tissue disorders) | 1 | 0
increased glare (Eye disorders) | 0 | 1
infection (Infections and infestations) | 2 | 0
cystitis (Renal and urinary disorders) | 1 | 0
left distal tibia/fibula fracture and surgery (Surgical and medical procedures) | 1 | 0
leg pain (both) (Musculoskeletal and connective tissue disorders) | 0 | 1
leukocytosis (Blood and lymphatic system disorders) | 1 | 0
low potassium (Blood and lymphatic system disorders) | 1 | 0
nausea (Gastrointestinal disorders) | 1 | 1
neck stiffness (Musculoskeletal and connective tissue disorders) | 0 | 1
peripheral retinopathy (PDR) (Eye disorders) | 1 | 0
neovascularization (Eye disorders) | 5 | 3
nocturnal leg cramps (Musculoskeletal and connective tissue disorders) | 0 | 1
ocular hypertension right eye (Eye disorders) | 0 | 1
oral surgery (Surgical and medical procedures) | 1 | 0
pain in right shoulder (Musculoskeletal and connective tissue disorders) | 0 | 1
purulent conjunctivitis (Eye disorders) | 1 | 0
pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
post-traumatic right shoulder adhesive capsulitis (Injury, poisoning and procedural complications) | 1 | 0
pre-retinal hemorrhage (Eye disorders) | 1 | 2
prostatitis (Renal and urinary disorders) | 0 | 1
pruritus during fluorescein angiography (Immune system disorders) | 1 | 0
punctate keratopathy (Eye disorders) | 1 | 0
received dentures (Product Issues) | 0 | 1
right ankle pain (Musculoskeletal and connective tissue disorders) | 0 | 1
right ankle sprain (Musculoskeletal and connective tissue disorders) | 1 | 0
right foot pain (Musculoskeletal and connective tissue disorders) | 0 | 1
right shoulder fracture (Injury, poisoning and procedural complications) | 1 | 0
shallow traction retinal detachment (Eye disorders) | 1 | 0
sinus infection (Respiratory, thoracic and mediastinal disorders) | 3 | 1
sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
sore throat (Infections and infestations) | 1 | 0
stomach virus (Infections and infestations) | 0 | 2
tendon release surgery (right hand) (Surgical and medical procedures) | 1 | 0
tendon release surgery (thumb) (Surgical and medical procedures) | 1 | 0
tooth extraction (Surgical and medical procedures) | 1 | 0
upper and lower teeth extracted (Surgical and medical procedures) | 0 | 1
upper respiratory infection (Respiratory, thoracic and mediastinal disorders) | 1 | 1
urinary retention (Renal and urinary disorders) | 0 | 1
urinary tract infection (Renal and urinary disorders) | 1 | 0
vertigo (Nervous system disorders) | 1 | 0
vitrectromy (Eye disorders) | 2 | 1
vitreous hemorrhage (Eye disorders) | 2 | 2

LIMITATIONS AND CAVEATS:
This is a proof of concept study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes